CLINICAL TRIAL: NCT04474769
Title: Supporting New Graduated Nurse's Professional Competence, a Theoretical Model for Optimal Orientation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Kirsi Lindfors, Pricipal Investigator, Tampere University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PreceptOR2014
Record Dates: First submitted 2020-06-28; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Competence; Nurse's Role

STUDY DESIGN:
Intervention Model Description: Longitudinal quasi-experimental intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention (Experimental): Intervention group's preceptors is given an eight-hour education entity about orientation and preceptorship. The objective is to enhance preceptors' knowledge and skills about the orientation and to give preceptors means to precept new graduate nurses better.
  Interventions: Other: Educational intervention for preceptors
- No intervention (No Intervention): Nursing units at the control group continue to precept as before.

INTERVENTIONS:
Other: Educational intervention for preceptors
  Arms: Educational intervention

SUMMARY:
This research is a longitudinal quasi-experimental intervention study which aim is to study education intervention's impact on new graduate nurses' orientation period, professional competence and organizational commitment. The study hypothesis is that new graduate nurses who start to work at the nursing unit which belong to the intervention group are more satisfied on received orientation, their professional competence develops faster and they are more committed to the organization than new graduate nurses at the units of the control group.

DETAILED DESCRIPTION:
This research is a dissertation which aim is to study nursing orientation from the preceptors' and new graduate nurses' point of view. The purpose is to develop a theoretical model for optimal orientation.

The aim is to study whether it is possible to affect new graduate nurses' professional competence development and their organizational commitment by educating preceptors. The aim is also to study new graduate nurses' perceptions of their clinical learning environment and received orientation and supporting and impeding factors of the successful orientation from the preceptors' point of view.

In order to measure the effectiveness of the education intervention on new graduate nurses' professional competence and commitment, participating nursing units is randomized by simple random sampling into the intervention group and the control group. Intervention group's preceptors is given an eight-hour education entity about orientation and preceptorship. The objective is to enhance preceptors' knowledge and skills about the orientation and to give preceptors means to precept new graduate nurses better. Nursing units at the control group continue to precept as before. The unit managers recruit participants (preceptors to the education intervention and new graduate nurses in both groups) to the study. No blinding has been made.

The independent variables are preceptors, work community, supervisors and new graduate nurses sociodemographic characteristics. The dependent variables are new graduate nurses' professional competence and commitment.

The data will be collected by using an electronical questionnaires. The Nurse Competence Scale (NCS©) will be used to study new graduate nurses' professional competence at the baseline, three months and nine months, a modified Clinical Learning Environment Scale (CLES+T©) will be used to study new graduate nurses' clinical learning environment and their orientation period at three months and Nurse Engagement Survey© will be used to study new graduate nurses' commitment at nine months. The same evaluations will be made in both groups. Preceptors' perceptions of the enhancing and impeding factors of the successful orientation is measured by open-ended questionnaire at the beginning of the education intervention.

The study results will be published on international nursing research journals and the theoretical model for optimal orientation will be published on doctoral dissertation.

ELIGIBILITY:
Inclusion Criteria:

* Less than one year from the graduation, willingness to participate

Exclusion Criteria:

* Already a registered nurse, more than one year from the graduation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Professional competence, the change of the professional competence is being assessed | Baseline
  Nurse Competence Scale, min 0 to max 100. Higher scores means better outcome
Professional competence, the change of the professional competence is being assessed | Three months
  Nurse Competence Scale, min 0 to max 100. Higher scores means better outcome
Professional competence, the change of the professional competence is being assessed | Nine months
  Nurse Competence Scale, min 0 to max 100. Higher scores means better outcome

SECONDARY OUTCOMES:
Precepting experience | Three months
  Clinical Learning Environment Scale, min 1 to max 10. Higher scores means better outcome
Organizational commitment | Nine months
  Nurse Engament Survey, min 1 to max 5. Higher scores means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Eija Paavilainen, PhD, Study Director — Tampere University

IPD SHARING:
Plan to Share IPD: No